CLINICAL TRIAL: NCT03533283
Title: An Open-Label, Multi-Center, Phase IB/II Study of Glofitamab and Atezolizumab or Polatuzumab Vedotin (Plus a Single Pre-Treatment Dose of Obinutuzumab) in Adult Patients With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: An Open-Label Phase lB/II Study of Glofitamab and Atezolizumab or Polatuzumab Vedotin in Adult Patients With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP39488
Record Dates: First submitted 2018-05-04; First posted 2018-05-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — glofitamab; atezolizumab; obinutuzumab; tocilizumab; polatuzumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atezolizumab (Experimental): Participants will receive Glofitamab in combination with Atezolizumab up to the maximum tolerated dose (MTD).
  Interventions: Drug: Glofitamab; Drug: Atezolizumab; Drug: Obinutuzumab; Drug: Tocilizumab
- Polatuzumab Vedotin (Experimental): Participants will receive Glofitamab in combination with polatuzumab vedotin up to the MTD.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab; Drug: Polatuzumab Vedotin
- Imaging Sub-study (Experimental): Participants will undergo positive-emission tomography/computed tomography (PET/CT) at screening, followed by an "Imaging Cycle," to replace Cycle 1 of the main study. Eligible participants will have the option roll-over to the atezolizumab arm of the main study from Cycle 2 onwards.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: 89Zr-Df-IAB22M2C

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered through IV infusion every 3 weeks (Q3W) beginning Cycle 1, Day 1, for up to 17 cycles (Cycle = 21 days). Step-up dosing, in which an initial lower dose will be followed by a higher dose 1 week later, will be considered for the initial treatment phase and for Cycle 9 of the re-treatment phase.
  Other Names: RO7082859; Columvi
Drug: Atezolizumab — Atezolizumab will be administered in combination with Glofitamab through IV infusion Q3W from Cycle 2, Day 1, for up to 16 cycles (Cycle = 21 days).
  Arms: Atezolizumab
Drug: Obinutuzumab — Obinutuzumab will be administered once, through IV infusion, at a fixed dose 7 days before the first dose of Glofitamab.
Drug: Tocilizumab — Tocilizumab will be administered as necessary to treat cytokine release syndrome (CRS).
  Other Names: Actemra
  Arms: Atezolizumab; Polatuzumab Vedotin
Drug: Polatuzumab Vedotin — Polatuzumab vedotin will be administered in combination with Glofitamab (on different days) Q3W from Cycle 1, Day 2, for up to 12 cycles (Cycle = 21 days).
  Arms: Polatuzumab Vedotin
Drug: 89Zr-Df-IAB22M2C — Participants will receive 89Zr-Df-IAB22M2C (Cycle 1 only) prior to obinutuzumab pre-treatment and again on Day 10 after dosing with glofitamab, followed by PET/CT.
  Arms: Imaging Sub-study

SUMMARY:
This is an open-label, single arm, multicenter, dose finding, Phase Ib study in order to assess the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) for this combination treatment and to evaluate the general safety, tolerability, pharmacokinetic (PK), pharmacodynamic, and preliminary anti-tumor activity of this combination treatment in adult patients.

This study includes an additional open-label imaging feasibility sub-study using a tracer in adult participants with relpased/refractory B-cell non-Hodgkin's lymphoma to image CD8+T-cells at baseline and after treatment with glofitamab, including pre-treatment with obinutuzumab.

ELIGIBILITY:
Main Inclusion Criteria

* Histologically-confirmed hematologic malignancy that is expected to express CD20 (Relapsed after or refractory to respond to at least one prior treatment regimen; no available treatment options that are expected to prolong survival or patients refusing chemotherapy or autologous stem cell transplant (SCT))
* Dose-escalation: Grades 1-3b relapsed or refractory (R/R) follicular lymphoma (FL) or marginal zone lymphoma (MZL) (nodal; extra-nodal; or splenic), diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), high-grade B-cell lymphoma (HGBCL) with MYC and BCL2 and/or BCL6 rearrangements (double-hit lymphoma), HGBCL not otherwise specified (NOS), DLBCL arising from FL (transformed FL)
* Dose-expansion: R/R LBCL, including DLBCL NOS, DLBCL arising from FL (transformed FL), PMBCL, HGBCL with MYC and BCL2 and/or BCL6 rearrangements (i.e., double-hit and triple-hit lymphomas), and HGBCL NOS
* At least one measurable target lesion
* Fresh pre-treatment biopsy, but if this cannot be taken, a previous archived biopsy from metastatic lesion can be taken as replacement if it is not older than 6 months and not confounded by major events (progression, treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ function (liver, hematological, renal)
* Negative test results for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV)

Inclusion Criteria Specific to Imaging Substudy

* At least two measurable target lesions
* Able to provide two fresh tumor biopsies (baseline and on-treatment)

Main Exclusion Criteria

* Participants with Chronic Lymphocytic Leukemia (CLL), acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma, Richter's transformation, CD20-positive ALL, Burkitt lymphoma, or lymphoplasmacytic lymphoma
* Current > Grade 1 peripheral neuropathy (only for participants being treated in the polatuzumab vedotin arm)
* Patients with known active infection, or reactivation of a latent infection within 4 weeks prior to Obinutuzumab (Gpt) infusion
* Patient with history of confirmed progressive multifocal leukoencephalopathy (PML)
* History of leptomeningeal disease
* Current or past history of central nervous system (CNS) lymphoma
* Current or past history of CNS disease
* Major surgery or significant traumatic injury </=28 days prior to Gpt infusion
* Significant cardiovascular disease or significant pulmonary disease
* Active or history of autoimmune disease or immune deficiency (with exceptions, e.g. hypothyroidism and Diabetes mellitus Type 1)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Treatment with any other standard anti-cancer radiotherapy / chemotherapy including investigational therapy within 4 weeks prior to Gpt infusion
* Prior solid organ transplantation
* Prior allogenic stem cell transplant (SCT)
* Autologous SCT within 100 days prior to Gpt infusion
* Documented refractoriness to an obinutuzumab-monotherapy regimen
* Prior treatment with anti-cancer/lymphoma therapies and systemic immunotherapeutic/immunostimulating agents within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to Gpt infusion
* Any history of immune related >/= Grade 3 adverse events (AE) with the exception of endocrinopathy managed with replacement therapy
* Ongoing corticosteroid use >25 milligrams/day of prednisone or equivalent within 4 weeks prior to and during study treatment
* Treatment with systemic immunosuppressive medication
* Administration of a live, attenuated vaccine within 4 weeks prior to Gpt infusion or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after last dose of study treatment

Exclusion Criteria Specific to Imaging Substudy

* Circulating lymphoma cells, defined by out of range (high) absolute lymphocyte count and/or the presence of abnormal/malignant cells in the peripheral blood differential signifying circulating lymphoma cell
* Participants who have had splenectomy or functional asplenia that could compromise protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Best Objective Response Rate (ORR) as Measured by Independent Review Committee (IRC) | Baseline until the end of treatment (13 to 14 months), then ever 3 months until end of study visit (to occur within 4 weeks of disease progression)
Dose Limiting Toxicities (DLTs) | Atezolizumab Arm: During DLT period of 21 days (or up to 42 days in the case of cycle delay), starting on Day 1, Cycle 2; Polatuzumab Vedotin Arm: During 5-week DLT period starting Cycle 1, Day 8

SECONDARY OUTCOMES:
Best ORR as Measured by Investigator | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Best Complete Response (CR) Rate, as Assessed by Fluorodeoxyglucose-Positron Emission Tomography/Computed Tomography (FDG-PET/CT) Scan | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Duration of Complete Response (DOCR) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Duration of Response (DOR) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Progression-Free Survival (PFS) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Event-Free Survival (EFS) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Time to First Complete Response (TFCR) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Time to First Overall Response (TFOR) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Overall Survival (OS) | Baseline through end of survival follow-up phase (survival follow-up is every 3 months until death, lost to follow-up, withdrawal of consent, or study termination)
Percentage of Participants with Adverse Events (AEs) | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Incidence and Severity of Cytokine Release Syndrome (CRS) Following Glofitamab Administration | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Anti-Drug Antibody (ADA) Formation | Baseline until end of treatment (13 to 14 months), then every 3 months until end of study visit (to occur within 4 weeks of disease progression)
Elimination Half-Life (T1/2) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Area Under the Concentration-Time Curve (AUC) for Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Time to Maximum Observed Serum Concentration (Tmax) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Maximum Observed Serum Concentration (Cmax) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Minimum Serum Concentration (Cmin) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Clearance (CL) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
Volume of Distribution at Steady-State (Vss) of Glofitamab Administered in Combination with Atezolizumab or Polatuzumab Vedotin | At pre-defined intervals through the end of study (EoS) visit (to occur within 4 weeks of disease progression)
CD8-Positive T Cell Proliferation | At pre-defined intervals during the study treatment period (up to 17 cycles; Cycle = 21 days)
CD20-Positive B-Cell Reduction | At pre-defined intervals during the study treatment period (up to 17 cycles; Cycle = 21 days)
SUVmax of 89Zr-Df-IAB22M2C (Imaging Sub-study) | From baseline to Day 13
SUVpeak of 89Zr-Df-IAB22M2C (Imaging Sub-study | From baseline to Day 13
SUVmean of 89Zr-Df-IAB22M2C (Imaging Sub-study) | From baseline to Day 13
Tumor Volume Based on 89Zr-Df-IAB22M2C PET-uptake (Imaging Sub-study) | From baseline to Day 13
Quantitation of CD8+ Cells on Biopsy Samples (Imaging Sub-study) | From baseline to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- UZ Gent, Ghent, Belgium
- Denmark (3):
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense C
- Israel (3):
  - Hadassah Ein Karem Hospital, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (4):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Asst Papa Giovanni Xxiii, Bergamo, Lombardy
  - Fond. IRCCS Istituto Nazionale Tumori, Milan, Lombardy
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - The HOPE Clinical Trials Unit, Leicester
  - University College London Hospitals NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Hutchings M, Sureda A, Bosch F, Larsen TS, Corradini P, Avigdor A, Terol MJ, Dominguez AR, Pinto A, Skarbnik A, Cordoba R, Jorgensen JM, Zinzani PL, Leung W, Bottos A, Li D, Relf J, Tandon M, Sellam G, Gritti G. Efficacy and Safety of Glofitamab Plus Polatuzumab Vedotin in Relapsed/Refractory Large B-Cell Lymphoma Including High-Grade B-Cell Lymphoma: Results From a Phase Ib/II Trial. J Clin Oncol. 2025 Dec 20;43(36):3788-3798. doi: 10.1200/JCO-25-00992. Epub 2025 Oct 20. PMID 41115257